CLINICAL TRIAL: NCT05637281
Title: Clinical Efficacy of Indomethacin in Early Treatment of Acute Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR2022467
Record Dates: First submitted 2022-11-15; First posted 2022-12-05 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2022-11

CONDITIONS: Acute Pancreatitis; Systemic Inflammatory Response Syndrome
Keywords: Non-steroidal anti-inflammatory drugs; indomethacin
MeSH Terms: conditions — Pancreatitis; Systemic Inflammatory Response Syndrome | interventions — Indomethacin; Congresses as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- convention (Placebo Comparator): patients in convention arm receive conventional management according to AP guidelines of International Association of Pancreatology and the Chinese Society of Gastroenterology, including goal-directed fluid resuscitation, oxygen supply even mechanical ventilation, and nutritional support if necessary.
  Interventions: Other: conventional treatment
- convention + indometacin (Experimental): Besides the conventional treatment,patients in convention + indometacin arm receive 50-mg indomethacin suppositories at intervals of 12 hours for a total of 6 doses.
  Interventions: Drug: Indometacin; Other: conventional treatment

INTERVENTIONS:
Drug: Indometacin — Besides the conventional treatment, indomethacin will be given to the patients in the convention + indomethacin group.
  Other Names: convention + indometacin
  Arms: convention + indometacin
Other: conventional treatment — All enrolled patients received conventional management according to AP guidelines of International Association of Pancreatology and the Chinese Society of Gastroenterology, including goal-directed fluid resuscitation, oxygen supply even mechanical ventilation, and nutritional support if necessary.
  Other Names: convention

SUMMARY:
Acute pancreatitis is a common critical disease of the digestive system. Accumulated data showed that overexpression of cyclooxygenase-2 (COX-2) in acute pancreatitis and experimental pancreatitis could be attenuated with COX-2 inhibitors. In recent years, it has been found that timely administration of indomethacin or diclofenac sodium to anus after ERCP can significantly reduce the incidence of AP after ERCP in patients at high risk of AP. The aim of this study was to evaluate the efficacy of rectal indomethacin in reducing the systemic inflammatory response syndrome (SIRS) score in AP patients.

ELIGIBILITY:
Inclusion Criteria:

(i) either gender aged 18-70 years; (ii) a confirmed diagnosis of AP; (iii) the time interval from the onset of symptoms to admission was no more than 48 h; (iv) written informed consent was obtained from the patients or their legal representatives.

Exclusion Criteria:

(i) pregnancy and breast feeding mother; (ii) severe chronic diseases such as cardiac dysfunction, chronic obstructive pulmonary disease, renal insufficiency, cirrhosis, inflammatory bowel diseases, and malignancies; (iii) peptic ulcer; (iv) pancreatitis due to trauma; (v) drug allergy; (vi) drug abuse and psychosis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2022-12-11 (Actual); Primary Completion 2023-12-11 (Estimated); Study Completion 2023-12-11 (Estimated)

PRIMARY OUTCOMES:
Systemic inflammatory response syndrome(SIRS) score at 72 hours after the initial intervention. | 72 hours after the initial intervention.
  The minimum value of SIRS is 0, and the maximum value of SIRS is 4. The higher score means a worse outcome.

SECONDARY OUTCOMES:
the serum levels of C-reactive protein(CRP) | 72 hours after the initial intervention.
  The normal range of CRP is 0-10mg/L, and the higher value means a worse outcome.
the serum levels of interleukin-6(IL-6) | 72 hours after the initial intervention.
  The normal range of IL-6 is 0-7pg/ml, and the higher value means a worse outcome.
score of abdominal pain | 72 hours after the initial intervention.
  The range of score of abdominal pain is 0-10, and the higher value means a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No